CLINICAL TRIAL: NCT04977895
Title: A Study to Assess Minimal Residual Disease by Next-generation Sequencing of Immunoglobulin Gene Rearrangements in Pediatric B-acute Lymphoblastic Leukemia
Brief Title: Monitoring Minimal Residual Disease（MRD）in Pediatric B-acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Professor, Sun Yat-sen University
Other Study IDs: MRD
Record Dates: First submitted 2021-07-11; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Minimal residual disease (MRD) monitoring — Minimal residual disease (MRD) assay using IgH-V(D)J NGS and FCM

SUMMARY:
This study aimed to investigate the performance of next-generation sequencing (NGS) techniques measuring immunoglobulin heavy chain (IgH)-variable, diversity, and joining (V[D]J) clonal rearrangements （IgH-V[D]J NGS） compared with flow cytometry (FCM) in detecting of minimal residual disease (MRD) for children with acute lymphoblastic leukemia treated with South Chinese Children Leukemia Group (SCCLG)-ALL 2016, and to predict the relapse of the disease in the early stage and to assess the prognosis, so as to provide the basis for early intervention treatment and reduce the hematological relapse and improve the survival rate.

DETAILED DESCRIPTION:
The measurement of residual leukemia levels, "minimal residual disease" (MRD), during therapy has now emerged as the most important predictor the outcome in acute lymphoblastic leukemia (ALL). As a result, risk-classifications based on MRD assessment has become an essential part of determining disease risk and directing therapeutic approach for children and adults with ALL.

Recently, next-generation sequencing (NGS) techniques measuring immunoglobulin (Ig) or T-cell receptor (TCR) clonal rearrangements as a method of detecting MRD have been introduced. These approaches expand the sensitivity of MRD detection to as high as 1 in 10,000,000 cells and have been shown to be predictive of relapse in children with ALL receiving standard chemotherapy.

In this study, the investigators will determine the sensitivity and specificity of IgH-V(D)J NGS and compared its capacity to measure MRD with that of flow cytometry using diagnostic and follow-up samples from more than 100 patients with ALL. Patients under age of 18 years with newly diagnosed ALL will be recruited and receive the treatment strategy of (SCCLG)-ALL 2016. After identifying a trackable clone in diagnostic samples (Baseline), MRD was measured using IgH-V(D)J NGS and FCM on bone marrow at 3 time-points: fifteen days after induction therapy (D15), thirty-three days after induction therapy (D33) and then at the end of induction therapy. Event-free survival (EFS), Relapse-free survival (RFS) and overall survival (OS) were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age≤18 years.
2. Newly diagnosed B-ALL.
3. No previous treatment.
4. Signed informed consent in keeping with the policies of the hospital.

Exclusion Criteria:

1. History of other malignancies, except in situ carcinoma or malignancy treated with curative intent.
2. Patients with active or uncontrollable infections such as hepatitis B, hepatitis C or HIV infection.
3. Patients with uncontrolled autoimmune diseases or immune defects. Other protocol-defined Inclusion/Exclusion may apply.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under age of 18 years with newly diagnosed B-ALL
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of MRD detection by IgH V(D)J NGS and FCM | During Induction Phase: up to 3 months
  The percentage of participants with MRD positive status from baseline to induction treatment completion determined by by IgH V(D)J NGS and FCM
Relapse-free survival (RFS) | up to 5 years
  RFS was estimated from the date of diagnosis until the date of relapse at any site. For other participants, last follow-up available was taken as last control. If participant did not complete study, date of last visit available was considered.

SECONDARY OUTCOMES:
MRD dynamic | During Induction Phase: up to 3 months
  MRD (IgH V(D)J NGS and/or FCM) dynamic between check-points
Overall survival (OS) | up to 5 years
  OS was defined as time from diagnostic date through the date of death due to any reasons. For all other participants, the last follow-up available was taken as the last control. If the participant had not completed the study, the date of the last visit available was considered.
Event-free survival (EFS) | up to 5 years
  EFS was estimated from date of diagnosis until date of one of the following events: relapse, refractory disease, second malignancy or death from any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Zhuo Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided